CLINICAL TRIAL: NCT06774092
Title: Prevalence of Anxiety Symptoms Among French General Practitioners
Acronym: Psy-MG
Status: Completed | Type: Observational
Sponsor: Université de Reims Champagne-Ardenne (Other)
Responsible Party: Sponsor
Other Study IDs: 2024_RIPH_02_Psy-MG
Record Dates: First submitted 2025-01-08; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Anxiety
Keywords: anxiety; self-employed GPs; prevalence
MeSH Terms: conditions — Anxiety Disorders | interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- GPs group: GPs, both qualified and established, practicing in France with at least some self-employed practice, who agreed to take part in the study.
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Data collection

SUMMARY:
Mental health is a major public health issue in the general population, but few studies seem to focus on the mental health of self-employed healthcare professionals, and GPs in particular. As front-line workers who are often called upon to manage complex situations, they are quite likely to suffer from anxiety-depressive symptoms or burnout. Nevertheless, general practice is vast, and there are many different ways of practising and organising it.

DETAILED DESCRIPTION:
The primary objective is to describe the prevalence of clinically significant anxiety symptoms in French self-employed GPs.

The secondary objective is to investigate the factors associated with the presence of clinically significant anxiety symptoms in French self-employed GPs.

ELIGIBILITY:
Inclusion Criteria:

* general practitioners
* qualified and established
* practicing in France
* with at least some self-employed practice
* agreeing to participate in the study

Exclusion Criteria:

* salaried general practitioners

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: GPs, both qualified and established, practicing in France with at least some self-employed practice, who agreed to take part in the study.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
anxiety | Day 0
  Anxiety will be evaluated using the Scale Trait Anxiety Inventory version Y (STAI-Y-A). The STAI Form Y-A consists of a set of twenty item sonly focus on the psychological and not the somatic aspects of anxiety. The STAI Form Y-A is a self-reported questionnaire. Each item is scored from 1 to 4 and a sum score of all items is computed. Higher score indicates greater anxiety. Presence of anxiety will be defined by a score greater than or equal to 46.

CONTACTS AND LOCATIONS:
Locations (1):
- Université de Reims Champagne Ardenne, Reims, France

IPD SHARING:
Plan to Share IPD: Undecided